CLINICAL TRIAL: NCT01902784
Title: Surrogate Project - Aim 2: Pilot Randomized Controlled Trial
Brief Title: The Surrogate Project (Surrogate Storytelling)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amber Barnato, MD, MPH, MS, Associate Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO13040209
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Surrogate Decision Maker, After Death of Patient
Keywords: Intensive Care Unit patients and families; Surrogate decision making; Life Sustaining Treatments (LST)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Storytelling Interview (Experimental): Participants assigned to receive the intervention will participate in an interview with a trained interventionist who will facilitate the telling of their 'story' - the personal experience they went through as a surrogate decision-maker for a loved one in the intensive care unit (ICU), who subsequently died after decisions were made to limit life-sustaining treatments (LST).
  These participants will be evaluated with questionnaires at baseline, 3 months, and 6 months after the death of their loved one (ICU patient).
  Interventions: Behavioral: Storytelling Interview
- Monitoring of well-being (No Intervention): Participants assigned to the Monitoring of well-being group will receive follow up phone calls from study staff and be evaluated with questionnaires at baseline, 3 months, and 6 months after the death of their loved one (ICU patient).

INTERVENTIONS:
Behavioral: Storytelling Interview
  Arms: Storytelling Interview

SUMMARY:
Research Protocol Abstract:

This is a phase II controlled trial (RCT) of a "storytelling" intervention compared to no treatment among surrogates who have participated in a decision to limit life-sustaining treatment in the ICU for an incapacitated loved one. Subjects will be sequentially assigned to "storytelling" (a facilitated elicitation of the experience 2-4 weeks after bereavement) or no treatment with follow up "monitoring of well-being". Subjects will receive print bereavement brochures at 1 week, and undergo telephone symptom assessment at 2-weeks, 3-months, and 6-months after bereavement.

ELIGIBILITY:
Inclusion Criteria:

Screening/Re-contact (1st phase)

* Eligible patients will:

  * lack decision-making capacity
  * have a surrogate decision maker (family member or friend)

Eligible surrogates will:

* be 18 years of age or older
* self-identify as having primary decision-making authority for the patient
* live within approximately 50miles or less of the University of Pittsburgh
* be able to conduct a 1hr interview in English

  * Court-appointed power of attorney will be excluded, as they are not expected to experience the same emotional distress as a family member or friend of a critically ill patient.

For Assignment to Intervention/Control (2nd phase)

* Eligible surrogates will:

  * have previously given consent for study staff to follow their loved one's course in the hospital and to be re-contacted
  * have participated in decision making about limitation of life-sustaining treatments (LST) for their loved one (ICU patient)
  * have had their loved one (ICU patient) die in the hospital

Exclusion Criteria:

Screening/Re-contact

* Ineligible patients will:

  * be less than 18 years old
  * prisoners
  * be of other legal concern, such as malpractice
* Ineligible surrogates will:

  * be less than 18 years old
  * be unable to complete a 1-hour interview and questionnaires in English
* For Assignment to Intervention/Control

Ineligible patients will:

* have fully and permanently regained decision-making capacity and therefore no longer require a surrogate to make treatment decisions
* be discharged from hospital alive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Acute referral to mental health services | 2-6 weeks after patient death (during or after participation in study intervention interview)
  We will assess acute risk of self-harm (or harm to others) and subsequent required referrals to mental health crisis services in participants throughout the intervention interview. Trained clinicians conducting interviews will refer when needed and record the number of participants requiring this service.
  Less than 5% of participants requiring an acute mental health crisis referral will be considered acceptable and an indicator of study safety.

SECONDARY OUTCOMES:
Research approach rates (participant interest) | start of recruitment - 6 months
  We will record the number of eligible surrogate decision makers who agree to be approached by a study staff member to hear about this research project, when asked by a member of their patient's clinical team. These counts will be summarized to assess a percentage and rate of eligible surrogates who agree to research approach among those who are eligible.
Randomization | 2- 6 weeks after patient death
  We will randomize participants who consent to participation in the 2nd portion of the study, after completion of a baseline questionnaire. Eligible participants will be randomized with equal numbers of participants in the intervention and control groups.
  Randomization of 30 eligible participants to the intervention group and 30 to the control will be considered successful and an indicator of study feasibility.
Experience of participation | 6 months (end of study participation)
  We will ask participants to report their experience of study participation by asking them, "How did participation in this study make you feel?" Five (5) answer choices will be given: Much better, Better, Neither better nor worse, Worse, or Much worse.
  10% or fewer participants reporting that the study made them feel 'Worse' or 'Much Worse' will be considered successful and an indicator of study acceptability.
Burdensomeness of participation | 6 months (end of study participation)
  We will ask participants to report how burdensome they felt participation in this study was for them by asking whether they Strongly Agree, Agree, Neither agree nor disagree, Disagree, or Strongly disagree with this statement: "Participating in this study was burdensome."
  10% or fewer participants reporting that the study was burdensome, with a response of 'Strongly Agree' or 'Agree' will be considered successful and an indicator of study acceptability.
Participation regret | 6 months (end of study participation)
  We will ask participants to report if they regret participation in this study by asking whether they Strongly Agree, Agree, Neither agree nor disagree, Disagree, or Strongly disagree with this statement: "I wish I hadn't agreed to participate in the study."
  10% or fewer participants reporting that they regret their participation in this study, with a response of 'Strongly Agree' or 'Agree' will be considered successful and an indicator of study acceptability.
enrollment rate | start of recruitment - end of study
  We will assess enrollment rate by recording the number of eligible participants who consent to participate and do participate in the intervention or control. The rate of enrollment will compare the number in this consented, participating group with the overall number of eligible participants encountered.
  We will consider an enrollment rate greater than 60% to be successful and an indicator of study feasibility.
completion of intervention session | 2 - 6 weeks after patient death
  We will record the number of eligible participants randomly assigned to the intervention session who complete the intervention session. We will calculate a rate of completion for the intervention session.
  A completion rate of 80% or greater will be considered successful and an indicator of study feasibility.
follow up questionnaire completion | 3 months +/- 9 days
  We will record the number of participants who complete the 3-month follow up questionnaire.
  A completion rate of 80% or greater will be considered successful and an indicator of study feasibility.
follow up questionnaire completion | 6 months +/- 18 days
  We will record the number of participants who complete the 6-month follow up questionnaire.
  A completion rate of 70% or greater will be considered successful and an indicator of study feasibility.

OTHER OUTCOMES:
Limit missing data | throughout study
  We will assess rates of missing data throughout data collection. A rate of 5% or lower missing data will be considered acceptable.
Participant distress after traumatic life event | 2-4 weeks after patient death (baseline questionnaire)
  We will summarize range and distribution of participant distress after a traumatic life event with the Impact of Events Scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant distress after traumatic life event | 3 months after patient death
  We will summarize range and distribution of participant distress after a traumatic life event with the Impact of Events Scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant distress after traumatic life event | 6 months after patient death
  We will summarize range and distribution of participant distress after a traumatic life event with the Impact of Events Scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant anxiety symptoms | 2-4 weeks after patient death (baseline questionnaire)
  We will summarize range and distribution of participant anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant anxiety symptoms | 3 months after patient death
  We will summarize range and distribution of participant anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant anxiety symptoms | 6 months after patient death
  We will summarize range and distribution of participant anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant depression symptoms | 2-4 weeks after patient death (baseline questionnaire)
  We will summarize range and distribution of participant depression symptoms with the Hospital Anxiety and Depression Scale (HADS) and the Primary Care Evaluation of Mental Disorders: Patient Health Questionnaire (PRIME-MD PHQ-9).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant depression symptoms | 3 months after patient death
  We will summarize range and distribution of participant depression symptoms with the Hospital Anxiety and Depression Scale (HADS) and the Primary Care Evaluation of Mental Disorders: Patient Health Questionnaire (PRIME-MD PHQ-9).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Participant depression symptoms | 6 months after patient death
  We will summarize range and distribution of participant depression symptoms with the Hospital Anxiety and Depression Scale (HADS) and the Primary Care Evaluation of Mental Disorders: Patient Health Questionnaire (PRIME-MD PHQ-9).
  Because this is a pilot trial, we will not conduct formal tests of efficacy.
Complicated grief symptoms | 6 months (+/- 3 weeks) after patient death
  We will assess whether surrogate participants are experiencing symptoms of complicated grief through administration of the Inventory of Complicated Grief during the final follow-up questionnaire at 6 months. Responses will be summarized to better understand how this population may be experiencing symptoms of complicated grief.
Subjective Units of Distress | 2-6 weeks after patient death (during & after completion of study intervention interview)
  We will ask participants to rate their present level of distress with the Subjective Units of Distress Scale (SUDS) based on a scale of 0-100, where 0 is absolutely calm and 100 is the worst distress imaginable, during and after their participation in the study intervention interview.
  Less than 20% of participants experiencing very high levels of distress (SUDS > 70) after the interview will be considered successful and an indicator of acceptable safety.
  Note: This is a projected level of acceptability with a subjective measure. Our multidisciplinary team will continue to evaluate the safety of participation throughout study.
Decision regret | 6 months (+/- 3 weeks) after patient death
  We will assess whether surrogate participants are experiencing regret over their decisions in the Intensive Care Unit (ICU) for their deceased loved one through administration of the Decision Regret Scale during the final follow-up questionnaire at 6 months. Responses will be summarized to better understand how this population may be experiencing symptoms of complicated grief.
Decision regret | 3 months (+/- 3 weeks) after patient death
  We will assess whether surrogate participants are experiencing regret over their decisions in the Intensive Care Unit (ICU) for their deceased loved one through administration of the Decision Regret Scale. Responses will be summarized to better understand how this population may be experiencing symptoms of complicated grief.
Decision regret | 2-4 weeks after patient death (baseline questionnaire)
  We will assess whether surrogate participants are experiencing regret over their decisions in the Intensive Care Unit (ICU) for their deceased loved one through administration of the Decision Regret Scale. Responses will be summarized to better understand how this population may be experiencing symptoms of complicated grief.

CONTACTS AND LOCATIONS:
Overall Officials: Amber E Barnato, MD MPH MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States